CLINICAL TRIAL: NCT01883167
Title: A Phase 1 Study to Evaluate the Potential Pharmacokinetic and Pharmacodynamic Interactions Between RDEA3170 and Febuxostat in Healthy Adult Male Subjects
Brief Title: RDEA3170 and Febuxostat Drug Interaction Study
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Ardea Biosciences, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: RDEA3170-105
Record Dates: First submitted 2013-06-18; First posted 2013-06-21 (Estimated); Last update posted 2014-01-09 (Estimated); Status verified 2014-01

CONDITIONS: Healthy
MeSH Terms: interventions — verinurad; Febuxostat

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Febuxostat (Experimental): Days 1-7: febuxostat 40 mg qd. Days 8-14: RDEA3170 10 mg or placebo qd in combination with febuxostat 40 mg qd.
  Days 15-21: RDEA3170 10 mg or placebo qd.
  Interventions: Drug: RDEA3170 10 mg; Drug: Febuxostat 40 mg; Drug: placebo
- RDEA3170 (Experimental): Days 1-7: RDEA3170 10 mg or placebo qd. Days 8-14: RDEA3170 10 mg or placebo qd in combination with febuxostat 40 mg qd.
  Days 15-21: febuxostat 40 mg qd.
  Interventions: Drug: RDEA3170 10 mg; Drug: Febuxostat 40 mg; Drug: placebo

INTERVENTIONS:
Drug: RDEA3170 10 mg — RDEA3170 10 mg once daily (qd)
Drug: Febuxostat 40 mg — Febuxostat 40 mg qd
Drug: placebo — placebo qd

SUMMARY:
This study will evaluate the potential pharmacokinetic (PK) and pharmacodynamic (PD) interaction between the XO inhibitor febuxostat and the investigational URAT1 inhibitor RDEA3170 and provide information for potential future clinical studies using this combination. Combination treatment using 2 drugs with different mechanisms of action may achieve improved response and may allow the use of lower doses, resulting in fewer side effects than the use of either drug alone.

ELIGIBILITY:
Inclusion Criteria:

* body weight ≥ 50 kg (110 lbs.) and a body mass index ≥ 18 and ≤ 40 kg/m2.
* no clinically relevant abnormalities in vital signs, ECG, physical examination or safety laboratory values, per the Investigator's judgment.
* a screening serum urate level ≥ 4.5 mg/dL.

Exclusion Criteria:

* history or suspicion of kidney stones.
* history of cardiac abnormalities as assessed during screening, including abnormal and clinically relevant electrocardiogram changes and/or family history of sudden death in otherwise healthy individual between the ages of 1 and 30 years.
* undergone major surgery within 3 months prior to Day 1.
* donated blood or experienced significant blood loss (> 450 mL) within 12 weeks prior to Day 1 or gave a plasma donation within 4 weeks prior to the Screening Period.
* inadequate venous access or unsuitable veins for repeated venipuncture.

Ages: 18 Years to 65 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2013-06; Primary Completion 2013-09 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
PK profile of RDEA3170 from plasma and urine and febuxostat from plasma | Days -1 (urine only), 7, 14, 21 and Days 8, 15, 22 (plasma only)
  Profile from plasma and urine in terms of AUC, Tmax, Cmax, t1/2, Ae, and CLr
  AUC: area under the concentration-time curve; Tmax: time to maximum plasma concentration; Cmax: maximum plasma drug concentration; t1/2: apparent terminal half-life; Ae: amount excreted of unchanged drug into urine; CLr: renal clearance

SECONDARY OUTCOMES:
PD profile of RDEA3170 and febuxostat alone and in combination | Days -1, 7, 14, 21 and Days 8, 15, 22 (serum only)
  Profile from serum and urine in terms of sUA concentration, renal clearance of uric acid, urine uric acid excretion amounts, and fractional excretion of uric acid.
  sUA: serum urate
Incidence of Adverse Events and Changes in Laboratory, Electrocardiogram, and Vital Signs Parameters | 8 weeks

CONTACTS AND LOCATIONS:
Overall Officials: S. Baumgartner, Study Director — Ardea Biosciences, Inc.
Locations (1):
- Kalamazoo, Michigan, United States

REFERENCES:
- [Derived] Rekic D, Johansson S, Leander J. Higher Febuxostat Exposure Observed in Asian Compared with Caucasian Subjects Independent of Bodyweight. Clin Pharmacokinet. 2021 Mar;60(3):319-328. doi: 10.1007/s40262-020-00943-6. Epub 2020 Sep 19. PMID 32951150